CLINICAL TRIAL: NCT02361879
Title: Ulipristal Acetate Versus GnRH Analogue Treatment Before Hysteroscopic Resection of Uterine Leiomyoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UPA and hysteroscopy
Record Dates: First submitted 2015-02-02; First posted 2015-02-12 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Fibroid
Keywords: fibroids; gnrh analogue; ulipristal acetate; hysteroscopy
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; Leuprolide

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulipristal acetate (Experimental): Womens will be treated with 5 mg/day of oral ulipristal acetate for 3 months
  Interventions: Drug: ulipristal acetate
- Leuprolile acetate (Active Comparator): women will be treated with 1 IM injection of leuprolide acetate 11,25 mg in in the luteal phase
  Interventions: Drug: Leuprolide acetate

INTERVENTIONS:
Drug: ulipristal acetate — 5 mg/day will be administered starting from day 1 of the cycle and up to three months later
  Other Names: Esmya
  Arms: Ulipristal acetate
Drug: Leuprolide acetate — One dose of 11.25 GnRH analogue depot will be administered in the luteal phase of the menstrual cycle (days 21-24)
  Other Names: Enantone 11.25
  Arms: Leuprolile acetate

SUMMARY:
The uterine leiomyoma is the most common female benign disease. Submucosal fibroid are about 10%, they distort the endometrial cavity causing heavy and/or irregular bleeding (AUB) and infertility. Hysteroscopic removal of submucosal myomas improves this conditions. GnRH analogues are commonly used before hysteroscopic myomectomy to make surgery easier and safer, but they are expensive, have potential side effects and lack a robust evidence base to support this practice. Ulipristal acetate treatment was able and faster to control in 90% of cases uterine bleeding associated with fibroids than GnRH agonists. UPA significantly improved quality of life and pain reduction.

DETAILED DESCRIPTION:
The uterine leiomyoma is the most common benign tumor of the female genital tract. The myomas are usually clinically apparent in 25% of patients. Submucosal fibroid are about 10% of all uterine myoma; they distort the endometrial cavity causing heavy and/or irregular bleeding (AUB) and infertility. According to the degree of myometrial penetration, the European Society for Gynaecological Endoscopy (ESGE) classified submucosal myomas in Type 0 (totally intracavitary fibroids), Type I (<50% myometral penetration), or Type II (>50% myometral penetration).

Hysteroscopic removal of submucosal myomas improves menorrhagia and AUB. GnRH analogues are commonly used before hysteroscopic myomectomy to make surgery easier and safer, but they are expensive, have potential side effects and lack a robust evidence base to support this practice. A recent meta-analysis of data demonstrated that symptomatic relief in patients undergoing surgery was similar either following pre-operative GnRH-a administration or without GnRH-a administration, mainly due to the persistence of abnormal bleeding due to the protrusion of the myoma into the uterine cavity.

In recent studies, Ulipristal acetate treatment was able to control uterine bleeding associated with fibroids in more than 90% of cases. Moreover, it controlled bleeding faster than GnRH agonists, with median times to amenorrhea of 5-7 days in patients receiving UPA compared to 21 days in patients receiving a GnRH agonist. It was demonstrated that UPA significantly improved also quality of life. Pain, as measured by the visual analogue scale, showed a degree of relief similar to that achieved for postoperative pain with narcotic and non-narcotic analgesics. This pain reduction is related to the high amenorrhea rate during treatment (severe bleeding being responsible for uterine contractions and prostaglandin secretion). No sub-analysis have been conducted on submucosal fibroids but, according to our experience, this subgroup of myomas may be the one who most benefits from the administration of UPA.

ELIGIBILITY:
Inclusion Criteria: submucosal leiomyoma, symptoms of menomethrorragia, menstrual disorder, infertility, pelvic pain.

Exclusion Criteria: intramural or subserosal leiomyomas, endometrial hyperplasia with atypia, history of uterine surgery

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Uterine bleeding assessed by pictorial blood-loss assessment chart (PBAC) | 90 days after the beginning of the treatment
  To compare the proportion of controlled uterine bleeding in patients with submucous myoma preoperatively treated by ulipristal acetate or by GnRh-a

SECONDARY OUTCOMES:
Feasibility of myoma hysteroscopic resection (VAS score) | Within 2 hours after the end of the hysteroscopy
  Surgeon experience about the hysteroscopy
Operative time | Within 2 hours after the end of the hysteroscopy
  It will be expressed in minutes
Haemoglobin concentration | The day before and 3 hours after the hysteroscopy
  It will be expressed in mg/dL
Fluid absorption | Within 2 hours after the end of the hysteroscopy
  It will be expressed in mL

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD,PhD, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, MD, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, Catanzaro, Italy